CLINICAL TRIAL: NCT06115811
Title: Development and Assessment of a Novel, Systematic Radiation Treatment Plan Evaluation Learning Tool for Radiation Oncology Residents
Brief Title: Radiation Treatment Plan Evaluation Learning Tool Pilot Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Beth Jimenez, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-021
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Radiation Oncology
Keywords: Radiation Oncology; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Treatment Plan Evaluation Learning Module (Experimental): Radiation oncology resident physicians will complete study procedures as below:
  * Initial survey and pre-module examination.
  * Learning module.
  * Post-module survey and examination.
  Interventions: Behavioral: Radiation Treatment Plan Evaluation Learning Tool

INTERVENTIONS:
Behavioral: Radiation Treatment Plan Evaluation Learning Tool — Web-based program comprised of a systematic, oncology treatment plan review system and learning modules. The case bank of radiation treatments plans is accessible via econtour.org.

SUMMARY:
This study involves both the development of a novel learning tool, the Radiation Treatment Plan Evaluation Learning Module, as well as a pilot program to validate this tool as an effective resource to teach treatment plan review and optimization to radiation oncology residents.

DETAILED DESCRIPTION:
This study involves both the development of a novel learning tool, the Radiation Treatment Plan Evaluation Learning Module, as well as a pilot program to validate this tool as an effective resource to teach treatment plan review and optimization to radiation oncology residents.

Stud procedures include screening for eligibility and completion of surveys and oncology examinations.

Participation is expected to last about 6-8 weeks.

It is expected about 20 radiation oncology resident physicians will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* The pilot program will be open to radiation oncology resident physicians that are in their PGY-2, PGY-3, or PGY-4 year.
* All residents must have completed a breast cancer-specific radiation oncology rotation at least 3 months prior to enrollment in the pilot program in order to be eligible.

Exclusion Criteria:

-The study will not include any special populations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Examination Score | Up to 8 weeks
  Analyzed with a paired samples t-test.

SECONDARY OUTCOMES:
Oncology Resident Confidence Rate | Week 1 - 8
  Scored using Likert scales and analyzed with non-parametric tests.
Oncology Resident Perceived Competence Rate | Week 1 - 8
  Scored using Likert scales and analyzed with non-parametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jimenez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation